CLINICAL TRIAL: NCT02201095
Title: Active Warming for Elective Caesarean Section - a RCT
Brief Title: Active Warming During Elective Caesearean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STH18196
Record Dates: First submitted 2014-07-15; First posted 2014-07-25 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Preoperative Hypothermia
Keywords: caesarean section; perioperative hypothermia; active warming; forced air warming; conduction mattress warming; thermal comfort; Prevention of

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal care (No Intervention): Normal care - no active warming
- Forced air warming (Active Comparator): Underbody forced air warming blanket
  Interventions: Device: Forced air warming
- Conduction warming mattress (Active Comparator): Underbody conduction warming mattress
  Interventions: Device: Conduction warming mattress

INTERVENTIONS:
Device: Forced air warming
  Other Names: Underbody bairhugger
  Arms: Forced air warming
Device: Conduction warming mattress
  Other Names: Inditherm conduction mattress
  Arms: Conduction warming mattress

SUMMARY:
During anaesthesia for caesarean section it is common to lose heat and become hypothermic, (<36 degrees C). In order to try and avoid this all women are given warmed intravenous fluid and insulated from cold surfaces. There are also 2 types of machine available to actively warm women;

1. Forced Air Warming - that uses a disposable sheet the woman lies upon with lots of air pockets that have warm air blown into them continuously by a fan.
2. Conduction Warming Mattress - a thin mattress which covers the operating table and the woman lies on top. The padded mattress has strips of material that heat up when electricity passes through it, similar to a normal electric blanket.

We plan to carry out a randomised controlled trial to compare these 2 methods with the current practice of no active warming.

The hypothesis for this study is that active warming women during elective caesarean section prevents women's temperature from dropping and keeps them more comfortable than if active warming were not used.

DETAILED DESCRIPTION:
When a baby is delivered by a surgical procedure (a caesarean section) the woman will usually have a "spinal" anaesthetic. With a "spinal", local anaesthetic is injected into the spinal fluid to make the woman numb from her chest to her feet, allowing her to be comfortable but awake during the birth. During this type of anaesthetic it is common to lose heat and become cold or "hypothermic" measured as less than 36 degrees Celsius. Becoming this cold can be uncomfortable for the woman but also causes other problems. It can make blood clotting less effective, alter the way wounds heal afterwards and make the woman more likely to develop infections or problems related to her heart and lungs.

To help keep their temperature stable, the investigators give all women fluid into the veins that is already warm and ensure that they are well insulated from any cold surfaces. There are two machines that the investigators can also use to actively warm patients but these are not yet used in every case. The first method is called "Forced Air Warming" and uses a special disposable sheet the woman lies upon with lots of air pockets that have warm air blown into them continuously by a fan. The woman is surrounded by these pockets of warm air, which help to warm her and also insulate against heat loss. The second method is called a "Conduction Warming Mattress" and uses a thin mattress which covers the operating table and the woman lies on top. The padded mattress has strips of material that heat up when electricity passes through it, similar to a normal electric blanket.

The investigators have already looked at the records of some women having caesarean sections in our hospital and found that both forced air warming and conduction mattress warming seem to help them stay warm. However, the investigators would like to study this in more detail and prove scientifically whether these methods are effective. Our aim in this study is to see if warming machines can help prevent women getting too cold, and prove scientifically whether one is more effective.

The hypothesis for this study is that active warming women during elective caesarean section prevents women's temperature from dropping and keeps them more comfortable than if active warming were not used.

The women will have exactly the same anaesthetic as they would have had if they were not in the study. If a woman agrees to be in the study she will be chosen randomly to receive either, normal care (including warmed fluids but no warming machines), additional warming with forced air or additional warming by conduction mattress. Her temperature will be measured at regular intervals before, during and after the caesarean section, at the same time she will be asked to score herself on a thermal comfort scale. The results will be analysed to compare the temperature changes in each group.

The investigators hope that the active warming machines will keep body temperature stable and prevent hypothermia. If the investigators find out that these machines prevent women getting cold, they can ensure that the most effective methods of warming during caesarean section operations are used and minimise problems due to becoming cold.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a singleton, uncomplicated pregnancy, presenting for elective caesarean section under spinal anaesthesia, where surgery and anaesthesia are expected to be uncomplicated. Patients scheduled for tubal ligation surgery (sterilisation) as part of the caesarean section may also be included.

Exclusion Criteria:

* Age under 18
* BMI <19 or >30
* Diseases of pregnancy: e.g. pregnancy induced hypertension
* Grand Multiparity - ie parity of 5 or greater
* Pre-operative pyrexia (temperature of 37.5 degrees C or greater)
* Pre-operative hypothermia (temperature 36.0 degrees or cooler)
* Significant co-existing maternal disease - e.g. congenital heart disease
* Co-existing maternal disease that could impact on temperature- e.g. hypo/hyperthyroid
* Coagulation abnormalities or anticipated excessive blood loss including any form of abnormal placentation
* Surgical procedure expected not to be routine/deviation from normal practice
* Condition preventing full, informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mean temperature on arrival in recovery | Temperature will be measured on arrival in recovery.
  The primary outcome of the study is to find whether there is a clinically significant statistical difference between the mean temperatures on arrival in recovery of the control and conduction mattress groups; the control and forced air warming groups; and the conduction mattress and forced air warming groups.

SECONDARY OUTCOMES:
Peri-operative hypothermia | Temperature will be measured evry 15 minutes throughout the duration of the procedure and in recovery room. The investigators anticipate that this will be over approximately a 2 hour period.
  To find whether these active warming devices significantly reduce the incidence of peri-operative hypothermia during spinal anaesthesia for caesarean section

OTHER OUTCOMES:
Thermal comfort scores | Thermal comfort will be assessed and scored at 15 minute intervals during surgery and in recovery. We anticipate that this will occur over approximately 2 hours.
  To assess whether active warming makes patients too hot and assess maternal thermal comfort and satisfaction during active warming.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Woolnough, Mb ChB, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Trust, Sheffield, South Yorkshire, United Kingdom